CLINICAL TRIAL: NCT03786367
Title: Mechanisms of Exertional Dyspnea in Chronic Thromboembolic Pulmonary Hypertension (CTEPH)
Brief Title: Dyspnea in Chronic Thromboembolic Pulmonary Hypertension
Status: Completed | Type: Observational
Sponsor: Dr. Denis O'Donnell (Other)
Collaborators: Queen's University (Other)
Responsible Party: Sponsor-Investigator, Dr. Denis O'Donnell, Principal Investigator, Queen's University
Organization: Queen's University (Other)
Other Study IDs: DMED-2208-18
Record Dates: First submitted 2018-11-15; First posted 2018-12-26 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension
Keywords: Dyspnea; Exertional Dyspnea; Pulmonary Hypertension; Exercise
MeSH Terms: conditions — Dyspnea; Hypertension, Pulmonary; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CTEPH: Clinically stable patients with Chronic Thromboembolic Pulmonary Hypertension (CTEPH) recruited from the Pulmonary Hypertension outpatient clinics at Hotel Dieu Hospital, Kingston, Ontario.
- Control: Age and sex-matched healthy control data collected as part of previous studies will be used as historic controls for this study.

SUMMARY:
Pulmonary embolism, or clots blocking the blood vessels of the lungs, is a common clinical condition requiring treatment with blood thinners. In most patients, recovery is complete. A small proportion of patients, however, develop complications (high blood pressure in the lung circulation, i.e. pulmonary hypertension). Persisting breathlessness during activity is a common symptom in many of these patients and leads to a reduced ability to engage in daily physical activity. The reason for this activity-related breathlessness remains uncertain and is the main question of the proposed study. Using new sophisticated technology, the investigators will determine the root causes of perceived breathing difficulty. The investigators will test the idea that breathlessness is fundamentally the result of increased drive to breathe from control centers in the brain. The investigators will measure drive to breathe by measuring the electrical activity descending from the brain to the main muscle of breathing - the diaphragm. The investigators will discover if the increased drive to breathe is due to accumulation of carbon dioxide in the blood as a result of poor blood perfusion of areas of the lung due to the effects of blockage by clots. The investigators also will investigate whether weakness and fatigue of the muscles of breathing, as a result of the high breathing demands that are present in patients with blood clots in the lungs, contribute to breathlessness. With this information it is hopeful that better treatment options will be developed to relieve this distressing symptom.

DETAILED DESCRIPTION:
Rationale: In patients with pulmonary embolism, most assessments of the burden of blood clots and possible related complications, currently rely on chest imaging and heart ultrasound. While these tests are useful in charting the course of the disease, they offer little about how the function of the heart and lungs is altered by the disease or the cause of common symptoms such as breathlessness during exercise. To better understand the reasons for persistent activity- related breathlessness in patients with a history of clots to the lungs, the investigators will undertake detailed assessment of breathlessness using validated scales and questionnaires during standardized exercise testing. At the same time the investigators will also measure a broad range of physiological tests that will indirectly measure how much blood perfusion of the lungs is reduced, how much the drive to breathe is increased, and whether there is additional strain and weakness of the muscles of breathing, particularly the diaphragm. This will allow the investigators to identify the main factors contributing to breathlessness in this population and will help to guide management. It is hoped that the development of simple new physiological markers or tests obtained during the stress of exercise can, in addition to conventional imaging, be used to monitor the course of the disease and response to treatment. In particular, the investigators hope that these new tests will help clinicians recognize at an early stage of the disease individuals more likely to develop progressive heart disease and breathing problems as a result of blood clots to the lungs.

Study design/methodology: This will be a single-centre, cross-sectional study observing the effect of Chronic Thromboembolic Pulmonary Hypertension (CTEPH) on exertional dyspnea and physiological responses to a standardized exercise task. After giving written informed consent, participants will complete 2 visits, each conducted in the morning 2-7 days apart. Visit 1 (screening for eligibility): medical history, symptom evaluation, complete pulmonary function testing, a symptom-limited incremental exercise test for familiarization of dyspnea assessments during exercise. Visits 2: pulmonary function testing (spirometry,) and a symptom-limited incremental exercise test to tolerance including detailed measurements of dyspnea (intensity, quality, affective dimensions), EMGdi and pressure-derived respiratory mechanical measurements. EMGdi will be used as an observational tool to measure inspiratory neural drive. An esophageal electrode-balloon catheter consisting of 5 electrode pairs will be inserted nasally and carefully positioned based on the strength of the EMGdi signal. EMGdi will be recorded continuously at rest and during exercise. The raw EMGdi signal will be sampled at 2000 Hz, band-pass filtered and converted to a root mean square (RMS) using computer software (LabChart). Maximal EMGdi (EMGdi,max) will be measured during inspiratory capacity (IC) maneuvers. EMGdi/EMGdi,max will be used as an index of the inspiratory neural drive to the crural diaphragm. Esophageal (Pes) and gastric pressures (Pga) will be recorded continuously at a rate of 200 Hz (PowerLab) using balloons mounted on the electrode catheter. Transdiaphragmatic pressure (Pdi) will be recorded as the difference between Pga and Pes signals. The continuous flow signal from the Vmax229d system will be input into the PowerLab system for offline analysis. Pre- and post-exercise inspiratory sniffs will be performed to obtain maximum Pes (Pes,sn) and Pdi (Pdi,sn). IC maneuvers at rest and throughout exercise will be used to obtain dynamic peak inspiratory Pes (Pes,IC) and Pdi (Pdi,IC). Pre- and post-exercise FVC maneuvers will also performed to obtain dynamic peak expiratory Pes (Pes,FVC). Respiratory mechanics will be analyzed as previously described (see reference). Vital signs will be monitored throughout exercise. Subjects will avoid caffeine, heavy meals, alcohol and major physical exertion prior to visits.

ELIGIBILITY:
Inclusion Criteria:

1. clinically stable as defined by stable hemodynamic status, optimized medical treatment, no changes in medication dosage or frequency of administration with no hospital admissions in the preceding 6 weeks
2. male or female ≥40 years of age
3. non-smoker
4. moderate-to-severe chronic activity-related dyspnea as defined by a modified Medical Research Council (MRC) dyspnea scale ≥2, or Baseline Dyspnea Index focal score ≤ 6
5. ability to perform all study procedures and provide/sign informed consent.

Exclusion Criteria:

1. women of childbearing age who are pregnant or trying to become pregnant
2. active cardiopulmonary disease or other comorbidities that could contribute to dyspnea and exercise limitation
3. important contraindications to clinical exercise testing, including inability to exercise because of neuromuscular or musculoskeletal disease(s)
4. use of daytime oxygen or exercise-induced O2 desaturation to < 80% on room air
5. body mass index (BMI) <18.5 or ≥35.0 kg/m2
6. other causes of significant pulmonary hypertension: pulmonary arterial hypertension, left heart disease, chronic pulmonary disease including, obstructive sleep apnea or pulmonary hypertension of unclear or multifactorial mechanism
7. systemic connective tissue disease

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will include 20 clinically stable patients with Chronic Thromboembolic Pulmonary Hypertension (CTEPH) recruited from the Pulmonary Hypertension outpatient clinics at Hotel Dieu Hospital, Kingston, Ontario.
  Healthy Control data will be from previous studies (no additional testing required in this group).
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Diaphragm electromyography (EMGdi) at a standardized time during cycle exercise test | Conducted at visit 2, 2-7 days after screening visit
  EMGdi will be used as an index of inspiratory neural drive. Assessments will be compared at a standardized time (at rest, during isotime and end-exercise) during incremental cycle ergometer exercise test.
Dyspnea intensity measured by the 10-point Borg Scale at a standardized time during cycle exercise test | Conducted at visit 2, 2-7 days after screening visit
  The 10-point Borg scale ranges from 0 "nothing at all" to 10 "maximal/extremely strong" and will be used to rate the intensity of dyspnea during exercise: a decrease in this rating signifies an improvement. Dyspnea intensity will be assessed at a standardized time (every minute) during incremental cycle ergometer exercise test.

SECONDARY OUTCOMES:
Inspiratory Capacity at a standardized time during cycle exercise test | Conducted at visit 2, 2-7 days after screening visit
  Exercise measurements of inspiratory capacity will be compared at a standardized time (at rest, during isotime and end-exercise) during incremental cycle ergometer exercise test.
Ventilation at a standardized time during cycle exercise test | Conducted at visit 2, 2-7 days after screening visit
  Exercise measurements of ventilation will be compared at a standardized time (at rest, during isotime and end-exercise) during incremental cycle ergometer exercise test.
Breathing frequency at a standardized time during cycle exercise test. | Conducted at visit 2, 2-7 days after screening visit
  Exercise measurements of breathing frequency (respiratory rate) will be compared at a standardized time (at rest, during isotime and end-exercise) during incremental cycle ergometer exercise test.
Carbon dioxide output (VCO2) at a standardized time during cycle exercise test. | Conducted at visit 2, 2-7 days after screening visit
  Exercise measurements of Carbon Dioxide output (VCO2) will be compared at a standardized time (at rest, during isotime and end-exercise) during incremental cycle ergometer exercise test.
Maximal oxygen uptake (VO2) at a standardized time during cycle exercise test. | Conducted at visit 2, 2-7 days after screening visit
  Exercise measurements of Maximal oxygen uptake (VO2) will be compared at a standardized time (at rest, during isotime and end-exercise) during incremental cycle ergometer exercise test.

CONTACTS AND LOCATIONS:
Overall Officials: Denis E O'Donnell, MD, Principal Investigator — Respiratory Investigation Unit, Queen's University
Locations (1):
- Respiratory Investigation Unit, Kingston General Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Faisal A, Alghamdi BJ, Ciavaglia CE, Elbehairy AF, Webb KA, Ora J, Neder JA, O'Donnell DE. Common Mechanisms of Dyspnea in Chronic Interstitial and Obstructive Lung Disorders. Am J Respir Crit Care Med. 2016 Feb 1;193(3):299-309. doi: 10.1164/rccm.201504-0841OC. PMID 26407036